CLINICAL TRIAL: NCT04477863
Title: Follow-up With Preimplantation Genetic Testing Patients
Status: Recruiting | Type: Observational
Sponsor: Genomic Prediction Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Genomic Prediction Inc 609
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Infertility; Genetic Disease; IVF
Keywords: PGT; Follow-up
MeSH Terms: conditions — Infertility; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Follow-up Interview — Non Applicable

SUMMARY:
The main purpose of this study is to perform longitudinal evaluations of clinical outcomes and personal perspectives following utilization of preimplantation genetic testing (PGT). Patients indicating willingness to participate in research during informed consent to perform PGT will be eligible for inclusion. A licensed genetic counselor will conduct a recorded interview.

DETAILED DESCRIPTION:
Purpose: To perform longitudinal studies of clinical outcomes and personal perspectives following utilization of PGT.

Background: Preimplantation Genetic Testing (PGT) is a commercially available adjunct to in vitro fertilization (IVF) and is now performed in over 40% of treatment cycles in the United Sates (Society for Assisted Reproductive Technology Annual Report, 2018). Several clinical genetics entities offer PGT services, including Genomic Prediction Clinical Laboratory (CLIA# 31D2152380, CAP# 8488628). It is common practice to perform interviews with, and record reviews of patients following clinical interventions. Results may provide instrumental information for the scientific and medical community to improve clinical care. We would like to review medical records in order to recruit patients to participate in longitudinal studies of clinical outcomes and personal perspectives following utilization of PGT.

Study Design and Methods: Patients indicating willingness to participate in research during informed consent to perform PGT will be eligible for inclusion. Patients who opted out of participating in research during informed consent to perform PGT will be ineligible for inclusion. Clinical PGT consent forms will be reviewed to identify patients that indicated willingness to participate in research. Eligible patients will be counseled on the study and consented for participation by a licensed genetic counselor. A total of 10,000 patients will be recruited. Following patient recruitment and informed consent, patient records and results of patient interviews may be used for publication in peer-reviewed scientific journals, presentation at scientific conferences or company meetings. As it is in standard practice, all external communication of results will maintain de-identification of all protected health information of all subjects (HIPAA guidelines). A licensed genetic counselor will conduct a recorded interview. Patient PGT, family history, and ethnicity data and information may be included in cohort analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicating willingness to participate in research during informed consent to perform PGT

Exclusion Criteria:

* Patients who opted out of participating in research during informed consent to perform PGT

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergo IVF and Preimplantation Genetic Testing
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-07-11 (Actual); Primary Completion 2050-07-11 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient perspectives on PGT | 2 years
  Analysis of interview responses

CONTACTS AND LOCATIONS:
Overall Officials: Nathan R Treff, PhD, Principal Investigator — Genomic Prediction
Locations (1):
- Genomic Prediction Clinical Laboratory, North Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Following patient recruitment and informed consent, patient records and results of patient interviews may be used for publication in peer-reviewed scientific journals, presentation at scientific conferences or company meetings.
Supporting Information: CSR
Time Frame: August 2020

REFERENCES:
- See also: SART Preliminary National Summary Report for 2018 — https://www.sartcorsonline.com/rptCSR_PublicMultYear.aspx?reportingYear=2018.